CLINICAL TRIAL: NCT00106314
Title: A Randomized, Double-Blind, Multi-Center, Dose Response, Efficacy and Safety Evaluation of Inflabloc Cap in the Treatment of Patients With Moderately Active Crohn's Disease
Brief Title: An Efficacy and Safety Evaluation of Inflabloc Cap in the Treatment of Patients With Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inflabloc Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL-C002-00
Record Dates: First submitted 2005-03-22; First posted 2005-03-23 (Estimated); Last update posted 2007-10-19 (Estimated); Status verified 2007-10

CONDITIONS: Crohn's Disease
Keywords: Dehydroepiandrosterone; DHEA; Crohn's disease; C-reactive protein; CRP; Crohn's Disease Activity Index; CDAI; Inflammatory Bowel Disease Questionnaire; IBDQ
MeSH Terms: conditions — Crohn Disease | interventions — Dehydroepiandrosterone

INTERVENTIONS:
Drug: Dehydroepiandrosterone [DHEA]

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Inflabloc Cap (Dehydroepiandrosterone [DHEA]) in the treatment of patients with moderately active Crohn's disease.

DETAILED DESCRIPTION:
This is a randomized, double-blind, multi-center, dose response, efficacy and safety study of Inflabloc Cap in patients with moderately active Crohn's disease. The primary objectives of the study are to evaluate the efficacy and safety of Inflabloc Cap in the treatment of patients with moderately active Crohn's disease who also have elevated CRP.

The study will be conducted at approximately 20 centers. Each patient will undergo screening followed by 8 weeks of treatment with Inflabloc Cap. Eligible male and female patients will be randomized in a 1:1:1 ratio to placebo, 30 mg, or 60 mg of DHEA administered twice daily via Inflabloc Cap so that approximately 60 patients complete the study. Following the Screening evaluations, consenting patients will self-administer 2 doses/day of study medication (placebo, 30 mg, or 60 mg of DHEA via Inflabloc Cap) for a total of 8 weeks (approximately 56 days). Patients will be required to complete a daily diary containing evaluations for number of liquid and soft stools, abdominal pain, fever and general well-being. Patients will also record use of study drug, concomitant medications and adverse events on the daily diary. Patients will be required to visit the study center at Screening, Baseline and at Weeks 1, 2, 4 and 8 following the initiation of treatment to turn in their diaries and any unused study medication, receive a physical exam and submit blood samples for chemistry, hematology and specialty laboratory measurements, and a urine sample for urinalysis. A stool sample is also required at Screening for culture and assay for C. difficile toxin. In addition, at the 8-week visit, patients will receive an exit exam including a physical exam (with ECG and vitals) and submit blood samples for chemistry, hematology and specialty laboratory measurements and a urine sample for urinalysis.

The primary efficacy endpoint for this study is defined as achieving a CDAI of 150 or less after 8 weeks of treatment. Secondary and exploratory efficacy endpoints at Weeks 4 and 8 will include achieving a CDAI of 150 or less (at 4 weeks), a change in CDAI from baseline of at least 100 points, a change from baseline in CRP, change from baseline in diarrhea and abdominal pain sub-scores, and change from baseline in IBDQ. Additionally, the safety of Inflabloc Cap when administered to patients with moderately active Crohn's disease with elevated CRP will be monitored through clinical evaluation, clinical laboratory data, collection of Adverse Events and other relevant safety evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Crohn's disease made at least 3 months prior to study entry.
* C-reactive protein above the upper limit of normal.
* Currently have moderately active Crohn's disease.

Exclusion Criteria:

* Women who are pregnant or lactating or of childbearing potential.
* History of colostomy, ileostomy, intestinal resection resulting in short bowel syndrome or symptomatic strictures.
* Symptoms (abdominal pain, vomiting) and radiographic evidence of mechanical bowel obstruction within the previous 6 months.
* Fistulizing disease.
* Positive stool culture for enteric pathogens and/or C. difficile toxin.
* History of significant disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2005-01; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Achieving CDAI (Crohn's Disease Activity Index) of 150 or less after 8 weeks of treatment

SECONDARY OUTCOMES:
Achieving a CDAI score of 150 or less at 4 weeks
Change in CDAI from baseline of at least 100 points at 4 and 8 weeks
Change in CRP (C-Reactive Protein) from baseline at 4 and 8 weeks
Change in health-related quality of life from baseline at 8 weeks as measured by the Inflammatory Bowel Disease Questionnaire (IBDQ)
Change from baseline in diarrhea and abdominal pain sub-scores from CDAI

CONTACTS AND LOCATIONS:
Overall Officials: Paul A. Litka, MD, Study Director — Inflabloc Pharmaceuticals, Inc.
Locations (38):
- United States (29):
  - Clinical Research Associates, Huntsville, Alabama
  - Advanced Clinical Research Institute, Anaheim, California
  - Sharp Rees-Stealy Medical Group, San Diego, California
  - Clinical Research of West Florida, Clearwater, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Northwest Gastroenterologists, Arlington Heights, Illinois
  - The University of Chicago Hospital, Chicago, Illinois
  - University of Louisville, Department of Internal Medicine, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Maryland Clinical Trials, Severna Park, Maryland
  - Jason Bodzin, MD, Farmington Hills, Michigan
  - AGA Clinical Research Associates, Egg Harbor, New Jersey
  - New York Center for Clinical Research, Lake Success, New York
  - Charlotte Gastroenterology and Hepatology, Charlotte, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Dept. of Gastroenterology, Cleveland, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Allegheny Center for Digestive Health, Pittsburgh, Pennsylvania
  - The Medical University of South Carolina, Charleston, South Carolina
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Atilla Ertan, MD, Houston, Texas
  - Mountain West Gastroenterology, Salt Lake City, Utah
  - SMG Reseach, Salt Lake City, Utah
  - University of Vermont College of Medicine / Fletcher Allen Health Care, Burlington, Vermont
  - McGuire DVAMC GI (111N), Richmond, Virginia
  - University of Washington Medical Center, Department of Gastroenterology, Seattle, Washington
  - Tacoma Digestive Disease Research Center, Tacoma, Washington
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin
- Canada (9):
  - GILDR Group, Edmonton, Alberta
  - Gastrointestinal Research Institute, Vancouver, British Columbia
  - Alan Cockeram, MD, Saint John, New Brunswick
  - IBD Clinical and Research Centre, Winnipeg, New Brunswick
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Doug Hemphill, MD, Barrie, Ontario
  - Credit Valley Digestive Disease Group, Mississauga, Ontario
  - Philip Hassard, MD, Ottawa, Ontario
  - Saskatoon Medical Specialists, Saskatoon, Saskatchewan

REFERENCES:
- [Background] Andus T, Klebl F, Rogler G, Bregenzer N, Scholmerich J, Straub RH. Patients with refractory Crohn's disease or ulcerative colitis respond to dehydroepiandrosterone: a pilot study. Aliment Pharmacol Ther. 2003 Feb;17(3):409-14. doi: 10.1046/j.1365-2036.2003.01433.x. PMID 12562454